CLINICAL TRIAL: NCT03468088
Title: The Relative Effect of Handgrip Strengthening Exercise in Treatment of the Patients With Primary Sub-Acromial Impingement Syndrome
Brief Title: Handgrip Strengthening Exercise in Treatment of the Patients With Primary Sub-Acromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Amal Alanazi, Post Graduate student, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAMS 039-3839
Record Dates: First submitted 2018-02-27; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Impingement Syndrome, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand grip strengthening (Experimental): This group will receive handgrip strengthening exercises.
  Interventions: Behavioral: Hand grip strengthening
- Conventional treatment (Active Comparator): This group will receive conventional exercises.
  Interventions: Behavioral: Conventional treatment

INTERVENTIONS:
Behavioral: Hand grip strengthening — Handgrip strengthening exercises will be added to the experimental group. This exercise is chosen based on literature review of EMG and biomechanical studies. Adjustable heavy grip hand gripper will be used as handgrip resistance at 10 repetitions maximum (RM). The exercise will be performed in standing position the patient's back will be rested in a wall, arm at 30º abduction, 60º abduction 90º abduction & with 90º ER. In this positions, the patient will be performed 3 sets of 10 squeezes each at a 1-minute interval.
  Arms: Hand grip strengthening
Behavioral: Conventional treatment — Ultrasound therapy will be used to treat both groups. Ultrasound will be applied; while the patient will be seated in an adjustable chair with back support, feet on the floor. The chair will be positioned beside a table. The patient's shoulder will be rested on the table beside the body and elbow will be flexed at 90°. A round-headed probe will be used that is put in direct contact with the patient's skin over the shoulder joint. Ultrasound gel will be used on all surfaces of the head in order to reduce friction and assist in the transmission of the ultrasonic waves.
  Arms: Conventional treatment

SUMMARY:
This study aims to investigate the relative effect of handgrip strengthening exercise in improving function, pain, strength, and active range of motion (AROM) of the shoulder among patients with primary sub-acromial impingement syndrome (SAIS).

DETAILED DESCRIPTION:
The current study is a Single-Blind Randomized Clinical Trial to investigate the effectiveness of handgrip strengthening exercise in the treatment of patients with primary subacromial impingement syndrome. The randomization process will be based on concealed envelop picked up by participants.The patient will be conveniently recruited from the ministry of health hospitals in Jeddah.The patient who will meet the inclusion criteria; they will sign the consent form. The baseline data will be collected. The assessment will be carried out at the baseline, 4 weeks and 8 weeks; end of the treatment program; by the same blinded examiner for each patient and consist of the following instrument: Disabilities of Arm, Shoulder & Hand (DASH questionnaire), Visual analog scale (VAS), Hand-held dynamometer (HHD), and smartphone clinometer.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with all study procedures and be available for the duration of the study
* Aged 18 to 45
* Diagnosed by their referring physician with subacromial impingement syndrome and has a positive impingement & rotator cuff test
* Pain intensity between 3 to 8 in VAS

Exclusion Criteria:

* History of shoulder fracture or dislocation, osteophytes, and labral tear.
* History of cardiac, neurological or musculoskeletal disease that precludes the ability to perform the exercise in the upper extremity.
* Treatment with another intervention.
* Hand or forearm dysfunction
* Rheumatoid disease
* Diabetic
* History of shoulder, cervical, and thoracic surgery
* Pregnancy
* Malignancy
* Symptoms for more than 1 year
* Bilateral SAIS

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Function | Change from baseline functional score at 8 weeks
  It will be assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, which is a 30-item questionnaire that assess the ability of a patient to perform various upper extremity activities. it uses a 5-point Likert scale. A higher scores signify a greater level of disability, whereas, lower scores signify a lower level of disability.

SECONDARY OUTCOMES:
Strength | Change from baseline muscle strength at 8 weeks
  It will be assessed using HHD
Range of motion | Change from baseline range of motion at 8 weeks
  It will be assessed using smartphone clinometer
Pain | Change from baseline pain intensity at 8 weeks
  Pain intensity will be assessed using visual analog scale (VAS) (0 - 10 cm with 0 indicates no pain and 10 indicates the worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Amal AlAnazi, Principal Investigator — King Saud University
Locations (1):
- Ministry of Health Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with the principal investigator (Ms. Amal AlAnazi) and sub-investigator (Dr. Ahmad Alghadir) due to confidentiality issues